CLINICAL TRIAL: NCT05860868
Title: Two Cycles VS Three Cycles Induction Chemotherapy Plus Concurrent Chemoradiotherapy in T1-4N2-3 Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Two Cycles VS Three Cycles Induction Chemotherapy in T1-4N2-3 Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Yong, Prof., First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Two VS Three
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 cycles (Experimental): 2 cycles induction + concurrent chemoradiotherapy
  Interventions: Drug: 2 cycles induction chemotherapy
- 3 cycles (Active Comparator): 3 cycles induction + concurrent chemoradiotherapy
  Interventions: Drug: 3 cycles induction chemotherapy

INTERVENTIONS:
Drug: 2 cycles induction chemotherapy — Drug: 2 cycles Induction Chemotherapy Induction regimens: TP (docetaxel 75 mg/m²; cisplatin 75 mg/m²) Q3w, TPF (docetaxel 60 mg/m²; cisplatin 60 mg/m²; 5-fluorouracil 600-750 mg/m² per day, continuous intravenous infusion d1-5) Q3w, or GP (gemcitabine: 1000 mg/m2 d1, d8; cisplatin 80 mg/m2) Q3w.
  Drug: Concurrent Chemotherapy Cisplatin 100 mg/m², Q3w.
  Radiation: Definitive Radiotherapy For all patients, the prescribed dose is 66-70 Gy (once a day, 5 times a week).
  Arms: 2 cycles
Drug: 3 cycles induction chemotherapy — Drug: 3 cycles Induction Chemotherapy Induction regimens: TP (docetaxel 75 mg/m²; cisplatin 75 mg/m²) Q3w, TPF (docetaxel 60 mg/m²; cisplatin 60 mg/m²; 5-fluorouracil 600-750 mg/m² per day, continuous intravenous infusion d1-5) Q3w, or GP (gemcitabine: 1000 mg/m2 d1, d8; cisplatin 80 mg/m2) Q3w.
  Drug: Concurrent Chemotherapy Cisplatin 100 mg/m², Q3w.
  Radiation: Definitive Radiotherapy For all patients, the prescribed dose is 66-70 Gy (once a day, 5 times a week).
  Arms: 3 cycles

SUMMARY:
This trial is a multi-center phase III clinical trial. The purpose of this trial is to explore whether 2 cycles induction chemotherapy combined with concurrent chemoradiotherapy is not inferior to 3 cycles induction chemotherapy combined with concurrent chemoradiotherapy in patients with locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Pathologically confirmed non-keratinizing nasopharyngeal carcinoma;
3. Stage T3-4N0-1 (according to the UICC/AJCC 8th);
4. No distant metastasis;
5. Have not received anti-cancer treatment in the past;
6. ECOG (Eastern Cooperative Oncology Group of the United States): 0-1;
7. Adequate hematologic, hepatic and renal function.

Exclusion Criteria:

1. The purpose of treatment is palliative;
2. Diagnosed with other malignant tumors at the same time;
3. Malignant tumor history;
4. Pregnancy or breastfeeding, or expect to become pregnant during the clinical trial period;
5. Combined serious illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
FFS, Failure Free Survival | 3 years
  Defined as the time from randomization to tumor recurrence, distant metastasis, or death due to any reason, whichever occurs first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: Undecided